CLINICAL TRIAL: NCT02181829
Title: Whole Lung IMRT in Children and Adults With Synovial Sarcoma and Lung Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-075
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2020-06

CONDITIONS: Synovial Sarcoma; Single or Multiple Lung Metastases
Keywords: Whole Lung IMRT; 14-075
MeSH Terms: conditions — Sarcoma, Synovial

ARMS (1):
- Whole Lung IMRT (Experimental): This is a single institution study involving patients with synovial sarcoma who have completed all standard therapy (e.g. surgery +/- radiation to the primary site) +/- any adjuvant chemotherapy. The sequence and types of therapy offered prior to WLI will likely vary based on primary tumor site, tumor resectability, extent of metastatic disease, performance status, and comorbidity. Each patient's therapy will be determined by the disease management team irrespective of participation on this protocol.
  Interventions: Radiation: Whole Lung IMRT

INTERVENTIONS:
Radiation: Whole Lung IMRT — External beam radiation therapy will be administered on an outpatient basis, once daily (except weekends and holidays) for approximately two weeks. Patients will undergo a simulation prior to initiation of radiation. Once an IMRT plan is generated which meets all dose constraints specified patients will be treated with 6MV photons for 10 treatments.

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, radiation has on the lungs has on the patient and on synovial sarcoma which has spread to the lungs. The standard treatment for synovial sarcoma which has spread to the lungs is chemotherapy with or without surgery to remove the tumors in the lungs. However, tumors often come back in the lungs after chemotherapy and/or surgery. Since synovial sarcoma is known to be sensitive to radiation, this study is looking at whether radiation therapy which is targeted to the entire lung can further reduce the chances of the cancer returning. This type of radiation is commonly used in other types of sarcoma to treat the cancer once it has spread to the lungs and it may be very useful in synovial sarcoma as well.

In this study, a special type of radiation will be used, called Intensity Modulated Radiation Therapy (IMRT). With IMRT the radiation beams are more customized to focus more radiation on the tumor cells while delivering less radiation to areas like the heart. The goal of this study is also to measure pulmonary toxicity and see if IMRT is feasible and has less toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with synovial sarcoma confirmed by MSKCC pathological review
* Patients with single or multiple lung metastases at diagnosis or that develop over the course of treatment. After completion of all chemotherapy, lung metastases or must be ≤ 2cm.
* Age ≥12 months of age
* Karnofsky performance status (KPS) must be ≥ 70 for patients ≥ 16 years of age and Lansky performance status must be ≥ 70 for patients < 16 years of age.
* Normal cardiac function
* No active coronary artery disease;
* No New York Heart Association class II, III or IV disease;
* No arrhythmia requiring treatment.
* Baseline echocardiogram with a shortening fraction of ≥27% or an ejection fraction ≥ 50%.
* Female patients of childbearing potential must have a negative pregnancy test within 14 days of radiation start.
* Female patients who are lactating must agree to stop breast-feeding.
* Sexually active patients of childbearing potential must agree to use effective contraception.

Exclusion Criteria:

* Patients with a history of prior radiation therapy to the thorax.
* Patients requiring a field size >40 cm as IMRT cannot be performed at extended SSDs.
* Patients with any concurrent medical or psychiatric condition or disease which, in the investigator's judgment, would make them inappropriate candidates for entry into this study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-07; Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Wolden, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Whole Lung IMRT
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Whole Lung IMRT
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 38 [23 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Evaluated for Toxicity
Description: The CTCAE version 4.0 scale will be used. The radiation oncologist will score toxicity at each visit.
Time Frame: within 3 months of the completion of treatment or 3 months following the completion of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Whole Lung IMRT
Number analyzed (Participants) | 10
Participants | 10

2. Secondary Outcome: Pulmonary Failure-free Survival
Description: A CT scan of the chest will be obtained. This study will use a modified Response Evaluation Criteria in Solid Tumor (RECIST) for assessment of tumor response. Pulmonary failure-free survival will be defined as survival with no progressive disease in the lungs.
Time Frame: pre-treatment, 3 and 6 months (+/- 3 weeks) and at 12, 18, and 24 months (+/- 6 weeks) post-treatment
Population: Data were not collected
Arm/Group | Whole Lung IMRT
Number analyzed (Participants) | 0

3. Secondary Outcome: Rates of Overall Survival (OS)
Description: Overall survival rates will be estimated by the Kaplan-Meier method.
Time Frame: two-year follow-up
Population: Data were not collected
Arm/Group | Whole Lung IMRT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months after first treatment
Arm/Group | Whole Lung IMRT
All-Cause Mortality (participants affected / at risk) | 7/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Whole Lung IMRT (N=10)
Nausea (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 4
Esophagitis (Gastrointestinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 1
Dysphagia (Gastrointestinal disorders) | 1
Platelet count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/29/NCT02181829/Prot_SAP_000.pdf